CLINICAL TRIAL: NCT02085863
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-way Crossover Drug-drug Interaction Study to Assess the Effect of Laquinimod 0.6 mg on the Pharmacokinetics and Pharmacodynamics of Ethinylestradiol and Levonorgestrel in Healthy Young Women
Brief Title: A Phase I Study in Young Healthy Women to Investigate the Effects of Laquinimod on Standard Oral Contraceptive When Both Treatments Are Given Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: TV5600-PK-10017; 2013-005356-14 (EudraCT Number)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laquinimod (Experimental): once daily oral doses of laquinimod (with combination oral contraceptives)
  Interventions: Drug: laquinimod; Drug: Placebo
- Placebo (Placebo Comparator): Matching placebo (with combination oral contraceptives)
  Interventions: Drug: laquinimod; Drug: Placebo

INTERVENTIONS:
Drug: laquinimod — Oral laquinimod 0.6 mg capsules (with oral contraceptives tablets containing 30 μg ethinylestradiol and 150 μg levonorgestrel (Microgynon®)
  Other Names: TV5600
Drug: Placebo — Placebo (with oral contraceptives tablets containing 30 μg ethinylestradiol and 150 μg levonorgestrel (Microgynon®)

SUMMARY:
This is a single center, randomized, double blind, placebo controlled, 2-way crossover drug-drug interaction (DDI) study to assess the effect of laquinimod on the PK and PD of ethinylestradiol (EE) and levonorgestrel (LNG) a commonly used oral contraceptive combination.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal women of age 18 to 40 years, who are healthy, non-pregnant and not planning pregnancy within the study period.
2. Women of childbearing potential who are willing to continuously use the oral contraceptive (OC) product containing EE 30 μg and LNG 150 μg from at least the commencement of their last normal period prior to the first dose of study medication and for a total of 4 consecutive cycles.
3. Willing to use a double barrier method of contraception (condom or diaphragm with spermicide) from screening until 30 days after the last laquinimod/placebo treatment. During administration of OC, the double barrier method should also be used.
4. Body Mass Index ranging from 18-30 kg/m2, inclusive.
5. Must be in a good health as determined by medical history, electrocardiogram (ECG), vital signs, physical and gynecological examination, and clinical laboratory tests.
6. Must have a regular menstrual cycle of 25 to 35 days (28-3/+7days) in the preceding 3 months prior to screening.
7. Subjects must be able to understand the requirements of the study and be willing to comply with the requirements of the study (eg, all dietary, exercise, tobacco and alcohol restrictions) and provide their written informed consent to participate in the study.

Exclusion Criteria:

1. Subjects who smoke at any frequency, have smoked in the last 6 months, or are planning to start smoking during the study, tobacco users, subjects currently using nicotine products (patches, gums, etc.) or subjects with a positive urine cotinine test at screening and/or at day -7.
2. Subjects with a known drug hypersensitivity to laquinimod, or one of its excipients (ie, mannitol, meglumine, or sodium stearyl fumarate).
3. Subjects with any significant food/drug allergies at the discretion of the investigator.
4. Subjects who are pregnant or lactating.
5. Subjects who had one of the following conditions in the noted amount of time prior to screening or at any time between screening and day -7: o Major trauma or surgery in the past 2 months.

   -Acute infection within 2 weeks (14 days).
6. Any malignancies, excluding basal cell carcinoma, prior to randomization.
7. Subjects who have any condition that possibly interferes with drug absorption, distribution, metabolism, or excretion.
8. Subjects suffering from, or with history of, one of the following: cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s), or a history of any illness that, in the opinion of the Investigator, might pose additional risk to the subject by participation in the study or confound the results of the study.
9. Subjects suffering from any condition in which the OC is contra indicated or not recommended.
10. Subjects who have used patches/intrauterine device/injectable hormonal contraception within 6 month prior to screening.
11. History of irregular menstruation.
12. Subjects with clinically relevant abnormality (judged by the investigator) of serum electrolytes or complete blood count.
13. Serum levels of ≥2× upper limit of normal alanine aminotransferase or aspartate aminotransferase or gamma-glutamyltransferase or alkaline phosphatase or direct bilirubin.
14. Subjects who have used one of the forbidden drugs or foods as following: o Excessive amounts (defined as daily intake of alcohol >40 g) of alcoholic beverages (eg, beer, wine, distilled spirits), or have a history of alcohol abuse, or are unwilling to comply with the restricted use of alcoholic beverages during the study.

    * An investigational drug (new chemical entity) during the 90 days or 5 half-lives prior to day -7 (whichever is longer).
    * Any medications, including over-the-counter medications or herbal preparations, used within 14 days prior to day -7 (except occasional paracetamol/acetaminophen or ibuprofen use and OC).
    * Any contraindicated concomitant medication according to the OC labeling.
    * Inducers or inhibitors of cytochrome P450 3A4 within 30 days prior to day -7.
    * Subjects who have consumed grapefruit, grapefruit juice, Seville oranges and pomelo-containing products, within the 14 days (2 weeks) prior to day -7.
15. Subjects with a positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, tetrahydrocannabinol) or positive test for ethanol at screening or at day -7.
16. Subjects who have donated or received any blood, plasma, or platelet transfusions in the 3 months prior to day -7, or who have made donations on more than 2 occasions within the 12 months preceding day -7, or who have planned donations during the study period or during the 3 months following the study.
17. Subjects with a positive screening test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody at screening.
18. Subjects who cannot participate or successfully complete the study, in the opinion of their general practitioner or the investigator, for the following reasons: o Subjects are under the legal age of consent or are mentally or legally incapacitated, or unable to give consent for any reason.

    * Subjects who are in custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitarium or social institution.
    * Subjects unable to be contacted in case of emergency.
    * Subjects who are employed by the Sponsor or the investigational site conducting the study
    * Any other reason, at the discretion of the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
AUC0-24 of EE and LNG plasma concentrations. | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
  to assess the effect of once daily oral doses of laquinimod on the pharmacokinetics (PK) of ethinylestradiol (EE) and levonorgestrel (LNG)
Cmax of EE and LNG plasma concentrations. | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
  to assess the effect of once daily oral doses of laquinimod on the pharmacokinetics (PK) of ethinylestradiol (EE) and levonorgestrel (LNG

SECONDARY OUTCOMES:
Tmax of EE and LNG plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Cmax of laquinimod plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
AUC0-24 of progesterone | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Ctrough of luteinizing hormone [LH], and follicle-stimulating hormone [FSH] | 10 min prior to dosing
Summary of Participants with Adverse Events | 25 Weeks
T1/2 of EE and LNG plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
CL/F of EE and LNG plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
V/F of EE and LNG plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Tmax of laquinimod plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
AUC0-24 of laquinimod plasma concentrations | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Cmax of progesterone | 10 min prior to dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 32415, Mönchengladbach, Germany